CLINICAL TRIAL: NCT00672958
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose Study Comparing the Efficacy and Safety of Lu AA21004 Versus Placebo in Acute Treatment of Adults With Major Depressive Disorder
Brief Title: Efficacy and Safety of Vortioxetine (Lu AA21004) in Treating Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LuAA21004_303; U1111-1114-2328 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Drug Therapy; Major Depressive Episode
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Vortioxetine placebo-matching capsules, orally, once daily for up to 6 weeks.
  Interventions: Drug: Placebo
- Vortioxetine (Experimental): Vortioxetine 5 mg, encapsulated tablet, orally, once daily for up to 6 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated immediate-release tablets.
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine
Drug: Placebo — Vortioxetine placebo-matching capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of once daily vortioxetine (Lu AA21004) in adults with major depressive disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called Vortioxetine. Vortioxetine is being tested to treat depression in adults who have major depressive disorder (MDD). This study looked at MDD relief in people who took vortioxetine.

The study enrolled 600 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 5 mg
* Placebo (dummy inactive pill) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in the United States. The overall time to participate in this study was approximately 94 days. Participants made 8 visits to the clinic, and were contacted by telephone 1 week, 2 weeks, and 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Suffers from a major depressive episode (MDE) as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria.
* The reported duration of the current MDE is at least 3 months.
* Has a Montgomery Åsberg Depression Rating Scale total score greater than or equal to 30.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Has received any investigational compound less than 30 days before Screening or 5 half-lives prior to Screening, whichever is longer.
* Has received Lu AA21004 in a previous clinical study.
* Has 1 or more the following:

  * Any current psychiatric disorder other than major depressive disorder as defined in the DSM-IV-TR (as assessed by the Mini International Neuropsychiatric Interview)
  * Current or past history of: manic or hypomanic episode, schizophrenia, or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
  * Any Axis II disorder that might compromise the study.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Narcotic analgesics
  * Nonsteroidal anti-inflammatory drugs
  * Rifampin
  * Macrolide antibiotics
  * Hormones (only thyroid hormone replacement, contraceptives [oral, patch], estrogen and progesterone replacement therapy are allowed in chronic use)
  * Hypoglycemic agents (chronic use is allowed)
  * Insulin (chronic use is allowed)
  * Systemic steroids
  * Quinidine
  * Antineoplastics
  * Antiobesity agents
* Has a significant risk of suicide according to the investigator's opinion or has a score greater than or equal to 5 on item 10 (suicidal thoughts) of the Montgomery Åsberg Depression Rating Scale or has made a suicide attempt in the previous 6 months.
* The current depressive symptoms are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each.
* Has received electroconvulsive therapy within 6 months prior to Screening.
* Is currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.
* Has a clinically significant unstable illness, for example, hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, infectious, skin and subcutaneous tissue disorders, or metabolic disturbance.
* Has an alanine aminotransferase, aspartate aminotransferase or total bilirubin level greater than 1.5 times the upper limits of normal.
* Has a serum creatinine greater than 1.5 times the upper limits of normal.
* Has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication. This criterion does not include basal cell or Stage I squamous cell carcinoma of the skin.
* Has clinically significant abnormal vital signs as determined by the investigator.
* Has an abnormal electrocardiogram determined by the central reader and confirmed as clinically significant by the investigator.
* Has 1 or more laboratory values outside the normal range, based on the blood or urine samples taken at the Screening Visit, that are considered by the investigator to be clinically significant.
* Has a thyroid stimulating hormone value outside the normal range at Screening Visit that is determined to be clinically significant by the investigator.
* Has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
* Has previously enrolled in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (33):
- United States (30):
  - Birmingham, Alabama
  - Cerritos, California
  - Encino, California
  - Fresno, California
  - San Diego, California
  - Farmington, Connecticut
  - Jacksonville, Florida
  - North Miami, Florida
  - Tampa, Florida
  - Hoffman Estate, Illinois
  - Lafayette, Indiana
  - Valparaiso, Indiana
  - Shreveport, Louisiana
  - Saint Paul, Minnesota
  - Florissant, Missouri
  - Saint Charles, Missouri
  - Las Vegas, Nevada
  - Rochester, New York
  - Dayton, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Lincoln, Rhode Island
  - North Charleston, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Lake Jackson, Texas
  - Wichita Falls, Texas
  - Brown Deer, Wisconsin
  - Middleton, Wisconsin
- Hull, Quebec, Canada
- Mexico (2):
  - Mexico City
  - San Luis Potosí City

REFERENCES:
- [Result] Jain R, Mahableshwarkar AR, Jacobsen PL, Chen Y, Thase ME. A randomized, double-blind, placebo-controlled 6-wk trial of the efficacy and tolerability of 5 mg vortioxetine in adults with major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):313-21. doi: 10.1017/S1461145712000727. Epub 2012 Sep 11. PMID 22963932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 47 investigative sites in the United States from 07 April 2008 to 12 November 2008.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 2 treatment groups, once a day placebo or 5 mg vortioxetine.
Groups:
- Vortioxetine: Vortioxetine 5 mg, encapsulated tablets, orally, once daily for up to 6 weeks.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine
Started | 300 | 300
Safety Set | 298 (All randomized patients who received at least 1 dose of double-blind study drug.) | 299 (All randomized patients who received at least 1 dose of double-blind study drug.)
Full Analysis Set | 286 (All safety set patients who had at least 1 valid postbaseline primary efficacy assessment.) | 292 (All safety set patients who had at least 1 valid postbaseline primary efficacy assessment.)
Completed | 236 | 244
Not Completed | 64 | 56
Not completed — Adverse Event | 11 | 9
Not completed — Lack of Efficacy | 6 | 11
Not completed — Non-compliance with study drug | 2 | 3
Not completed — Protocol deviations | 11 | 5
Not completed — Voluntary withdrawal | 12 | 8
Not completed — Lost to Follow-up | 22 | 17
Not completed — Reason not specified | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine | Total
Number analyzed (Participants) | 300 | 300 | 600
Age Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.70) | 42.5 (13.04) | 42.4 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 186 | 350
  Male | 136 | 114 | 250
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White, including Hispanic) | 216 | 209 | 425
  Black | 78 | 81 | 159
  Asian | 4 | 8 | 12
  American Indian or Alaska Native | 2 | 1 | 3
  Native Hawaiian/ Other Pacific Islander | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 36 | 34 | 70
  Non-Hispanic/Non-Latino | 264 | 266 | 530
Region of Enrollment [Number; unit: participants]
  United States | 300 | 300 | 600
Weight [Mean (Standard Deviation); unit: kg] | 89.53 (23.326) | 86.63 (23.528) | 88.08 (23.453)
Height [Mean (Standard Deviation); unit: cm] | 170.36 (9.815) | 168.67 (9.815) | 169.51 (9.843)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.84 (7.675) | 30.48 (8.217) | 30.66 (7.946)
Waist circumference [Mean (Standard Deviation); unit: cm] | 97.58 (17.757) | 96.22 (18.961) | 96.90 (18.366)
Smoking classification [Number; unit: participants]
  Never smoked | 119 | 123 | 242
  Current smoker | 124 | 116 | 240
  Ex-smoker | 57 | 61 | 118
Alcohol consumption [Number; unit: participants]
  Never | 108 | 106 | 214
  Once monthly or less often | 102 | 124 | 226
  Once per week | 46 | 41 | 87
  2-to-6 times/week | 33 | 21 | 54
  Daily | 11 | 8 | 19
24-item Hamilton Depression Scale total score [Mean (Standard Deviation); unit: scores on a scale] — The 24-item Hamilton Depression Scale (HAM-D24) is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74, where a higher score indicates a greater depressive state.
  scores on a scale | 32.2 (5.50) | 32.7 (5.42) | 32.5 (5.46)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 34.0 (3.41) | 34.1 (3.39) | 34.1 (3.40)
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety.
  scores on a scale | 19.5 (6.19) | 19.3 (5.24) | 19.4 (5.73)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.8 (0.66) | 4.8 (0.68) | 4.8 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-item Hamilton Depression Scale Total Score at Week 6
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score range is from 0 to 74 where a higher score indicates a greater depressive state. Least squares (LS) means were from an Analysis of Covariance (ANCOVA) model with treatment and center as fixed factors and the baseline value as a covariate.
Time Frame: Baseline and Week 6
Population: The full analysis set, which includes all randomized participants who received at least 1 dose of study drug and had at least 1 postbaseline value for assessment of primary efficacy. Last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
scores on a scale | -13.87 (0.662) | -14.61 (0.650)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine; Change from Baseline in HAM-D24 total score at Week 6 was tested at significance level 0.05. To control for multiplicity, subsequent endpoints were to be tested in a sequential testing procedure at significance level 0.025; as soon as an endpoint in a sequence was non-significant at 0.025, the testing procedure was stopped for all subsequent endpoints in that sequence; Test type: Superiority or Other; p = 0.407, ANCOVA — Pre-specified sequential statistical testing procedure indicates that when p-value for change from baseline in HAMD-24 at Week 6 >0.05, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; Analysis of covariance (ANCOVA), with treatment and center as fixed factors and baseline HAM-D24 as a covariate; LS Mean Difference = -0.74, 95% CI 2-sided [-2.48 to 1.01]

2. Primary Outcome: Change From Baseline in the 24-item Hamilton Depression Scale Total Score at Other Weeks Assessed
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74 where a higher score indicates a greater depressive state. LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 3, 4 and 5
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
scores on a scale
  Week 1 (n=281, 286) | -6.03 (0.394) | -5.96 (0.387)
  Week 2 (n= 286, 291) | -9.30 (0.505) | -9.05 (0.496)
  Week 3 (n= 286, 292) | -11.05 (0.545) | -11.73 (0.536)
  Week 4 (n= 286, 292) | -12.33 (0.579) | -12.66 (0.568)
  Week 5 (n=286, 292) | -13.11 (0.628) | -13.98 (0.617)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine; Comparison of change from Baseline at Week 1; Test type: Superiority or Other; p = 0.901, ANCOVA; ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS Mean Difference = 0.07, 95% CI 2-sided [-0.97 to 1.10]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine; Change from Baseline at Week 2; Test type: Superiority or Other; p = 0.701, ANCOVA; ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS Mean Difference = 0.26, 95% CI 2-sided [-1.07 to 1.59]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine; Change from Baseline at Week 3; Test type: Superiority or Other; p = 0.356, ANCOVA; ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS Mean Difference = -0.68, 95% CI 2-sided [-2.11 to 0.76]
Statistical Analysis 4: Comparison: Placebo vs Vortioxetine; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.670, ANCOVA; ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS Mean Difference = -0.33, 95% CI 2-sided [-1.85 to 1.19]
Statistical Analysis 5: Comparison: Placebo vs Vortioxetine; Change from Baseline at Week 5; Test type: Superiority or Other; p = 0.304, ANCOVA; ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS Mean Difference = -0.87, 95% CI 2-sided [-2.52 to 0.79]

3. Secondary Outcome: Percentage of Responders in HAM-D24 Total Score by Study Visit
Description: A responder is defined as a participant with a ≥50% decrease from Baseline in HAM-D24 total score. The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74, where a higher score indicates a greater depressive state.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5 and 6.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
percentage of participants
  Week 1 (n=281, 286) | 7.8 | 7.0
  Week 2 (n=286, 291) | 23.8 | 21.0
  Week 3 (n=286, 292) | 31.8 | 32.9
  Week 4 (n=286, 292) | 39.2 | 37.0
  Week 5 (n=286, 292) | 44.4 | 43.8
  Week 6 (n=286, 292) | 46.2 | 46.2

4. Secondary Outcome: Percentage of Participants in MADRS Remission at Week 6
Description: Remission is defined as a participant with a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≤10. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Week 6
Population: Full analysis set; LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
percentage of participants | 32.2 | 29.1

5. Secondary Outcome: Percentage of Participants With a Sustained Response in HAM-D24
Description: A sustained response is defined as a ≥20% decrease from Baseline in HAM-D24 total score obtained at Week 1 and sustained through Week 5 and at least 50% decrease from Baseline at Week 6.
Time Frame: Baseline to Week 6
Population: Full analysis set. Participants with missing values were classified as nonsustained responders/remitters.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
percentage of participants | 21.0 | 19.5

6. Secondary Outcome: Change From Baseline in Montgomery Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. Least square means are from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5 and 6.
Population: Full analysis set. LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
scores on a scale
  Week 1 (n=281, 286) | -6.88 (0.418) | -6.38 (0.412)
  Week 2 (n=286, 291) | -10.57 (0.530) | -9.82 (0.523)
  Week 3 (n=286, 292) | -12.48 (0.583) | -12.76 (0.575)
  Week 4 (n=286, 292) | -13.72 (0.624) | -13.70 (0.615)
  Week 5 (n=286, 292) | -14.40 (0.673) | -15.12 (0.664)
  Week 6 (n=286, 292) | -15.48 (0.708) | -15.80 (0.698)

7. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A)
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. Least squares means are from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4 and 6.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
scores on a scale
  Week 1 (n=281, 286) | -3.25 (0.288) | -3.21 (0.284)
  Week 2 (n=286, 291) | -4.92 (0.343) | -4.77 (0.338)
  Week 4 (n=286, 292) | -6.52 (0.393) | -6.88 (0.387)
  Week 6 (n=286, 292) | -7.60 (0.419) | -7.84 (0.413)

8. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity of Illness
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5 and 6.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
scores on a scale
  Week 1 (n=281, 286) | -0.47 (0.045) | -0.40 (0.044)
  Week 2 (n=286, 291) | -0.82 (0.061) | -0.82 (0.060)
  Week 3 (n=286, 292) | -1.07 (0.069) | -1.08 (0.067)
  Week 4 (n=286, 292) | -1.25 (0.073) | -1.20 (0.072)
  Week 5 (n=286, 292) | -1.28 (0.079) | -1.36 (0.077)
  Week 6 (n=286, 292) | -1.46 (0.085) | -1.46 (0.083)

9. Secondary Outcome: Clinical Global Impression Scale-Global Improvement Scale
Description: The Clinical Global Impression - Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from an ANCOVA model with treatment and center as fixed factors and the CGI-S Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5 and 6.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
scores on a scale
  Week 1 (n=281, 286) | 3.38 (0.048) | 3.46 (0.047)
  Week 2 (n=286, 291) | 3.09 (0.062) | 3.08 (0.061)
  Week 3 (n=286, 292) | 2.90 (0.066) | 2.84 (0.065)
  Week 4 (n=286, 292) | 2.74 (0.070) | 2.75 (0.069)
  Week 5 (n=286, 292) | 2.74 (0.073) | 2.65 (0.071)
  Week 6 (n=286, 292) | 2.61 (0.076) | 2.57 (0.075)

10. Secondary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale - Self-assessment (MADRS-S)
Description: The MADRS-S is a patient-reported outcome measure based on MADRS, administered to evaluate treatment effectiveness in depression. This scale consists of 9 items assessing patients' mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life. Each item is scored between 0 (best) and 3 (worst). The total score is calculated by summing the answers of the nine items, ranging between 0 and 27 (higher scores indicate increased impairment). LS means are from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Weeks 1, 4 and 6.
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
scores on a scale
  Week 1 (n=279, 286) | -2.81 (0.214) | -2.73 (0.210)
  Week 4 (n=284, 292) | -4.18 (0.272) | -4.05 (0.267)
  Week 6 (n=284, 292) | -4.56 (0.313) | -4.97 (0.307)

11. Secondary Outcome: Change From Baseline in 36-item Short-form Health Survey (SF-36) at Week 6
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The 8 health concepts are: 1. Limitation in physical activities because of health problems. 2. Limitations in usual role activities because of physical health problems. 3. Bodily pain. 4. Limitations in social activities because of physical or emotional problems. 5. General mental health (psychological distress and well-being). 6. Limitations in usual role activities because of emotional problems. 7. Vitality (energy and fatigue). 8. General health perception. Each scale ranges from 0 (best) - 100 (worst). LS means are from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 6
Population: Full analysis set where Baseline SF-36 data were available; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 279 | 287
scores on a scale
  Physical functioning | 5.47 (1.277) | 6.87 (1.264)
  Role - physical | 11.73 (1.569) | 14.41 (1.549)
  Bodily pain | 10.77 (1.460) | 10.39 (1.445)
  General health | 7.65 (0.985) | 7.37 (0.975)
  Vitality | 18.00 (1.455) | 17.34 (1.440)
  Social functioning | 21.34 (1.687) | 22.01 (1.667)
  Role - emotional | 19.43 (1.756) | 20.76 (1.732)
  Mental health | 18.98 (1.401) | 20.00 (1.385)

12. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 6
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from an ANCOVA model with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 6
Population: Full analysis set where data were available; LOCF was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 217 | 220
scores on a scale | -6.61 (0.548) | -6.69 (0.557)

13. Secondary Outcome: Health Care Resource Utilization as Assessed by the Health Economic Assessment Questionnaire
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors the participants absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 6
Population: Full analysis set.
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine
Number analyzed (Participants) | 286 | 292
participants
  Baseline: Any resource use | 82 | 77
  Baseline: Any hospitalization-related services | 1 | 0
  Baseline: Hospitalization related to depression | 1 | 0
  Baseline: Any sick leave | 16 | 21
  Baseline: Sick leave related to depression | 9 | 13
  Week 6: Any resource use | 58 | 41
  Week 6: Any hospitalization-related service | 3 | 1
  Week 6: Hospitalization related to depression | 0 | 0
  Week 6: Any sick leave | 7 | 7
  Week 6: Sick leave related to depression | 3 | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are defined as adverse events whose onset occurred or intensity increased after the first dose of double-blind study drug through 30 days after permanent discontinuation of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine
Serious Adverse Events (participants affected / at risk) | 4/298 | 7/299
Other Adverse Events (participants affected / at risk) | 142/298 | 168/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=298) | Vortioxetine (N=299)
Drug hypersensitivity (Immune system disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Puncture site infection (Infections and infestations) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=298) | Vortioxetine (N=299)
Nausea (Gastrointestinal disorders) | 28 | 57
Diarrhoea (Gastrointestinal disorders) | 21 | 34
Dry mouth (Gastrointestinal disorders) | 19 | 25
Abdominal pain (Gastrointestinal disorders) | 3 | 12
Dyspepsia (Gastrointestinal disorders) | 10 | 5
Constipation (Gastrointestinal disorders) | 6 | 9
Vomiting (Gastrointestinal disorders) | 4 | 8
Fatigue (General disorders) | 7 | 5
Irritability (General disorders) | 7 | 3
Nasopharyngitis (Infections and infestations) | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Urinary tract infection (Infections and infestations) | 5 | 6
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Headache (Nervous system disorders) | 45 | 51
Dizziness (Nervous system disorders) | 22 | 19
Somnolence (Nervous system disorders) | 10 | 11
Insomnia (Psychiatric disorders) | 9 | 6
Depression (Psychiatric disorders) | 5 | 7
Initial insomnia (Psychiatric disorders) | 4 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.